CLINICAL TRIAL: NCT04614948
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study to Assess the Efficacy and Safety of Ad26.COV2.S for the Prevention of SARS-CoV-2-mediated COVID-19 in Adults Aged 18 Years and Older
Brief Title: A Study of Ad26.COV2.S for the Prevention of SARS-CoV-2-mediated COVID-19 in Adults
Acronym: ENSEMBLE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108916; 2020-003643-29 (EudraCT Number); VAC31518COV3009 (Other: Janssen Vaccines & Prevention B.V.)
Expanded Access: NCT04817657 (No longer available)
Record Dates: First submitted 2020-11-03; First posted 2020-11-04 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Participants With or Without Stable Co-morbidities Associated With Progression to Severe COVID-19
MeSH Terms: interventions — Ad26COVS1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ad26.COV2.S (Experimental): Participants will receive intramuscular (IM) injection of Ad26.COV2.S vaccine on Day 1 and Day 57 in the double-blind phase. At unblinding visit (open-label phase), participants who have not yet received second vaccination will receive second dose of Ad26.COV2.S vaccine on Day 57, if applicable and newly enrolled participants will either receive IM injection of one dose of Ad26.COV2.S vaccine on Day 1 or two doses of Ad26.COV2.S vaccine on Day 1 and Day 57. All ongoing participants who only received a single vaccination with Ad26.COV2.S in the study will be offered to receive single booster dose of Ad26.COV2.S in the open label phase preferably within 6 to 12 months after the participant's first Ad26.COV2.S vaccination.
  Interventions: Biological: Ad26.COV2.S
- Placebo (Placebo Comparator): Participants will receive IM injection of placebo on Day 1 and Day 57 in the double-blind phase. At unblinding visit (open-label phase), participants initially receiving placebo will be offered to receive IM injection of a single dose of Ad26.COV2.S vaccine. All ongoing participants who only received a single vaccination with Ad26.COV2.S in the study will be offered to receive single booster dose of Ad26.COV2.S in the open label phase preferably within 6 to 12 months after the participant's first Ad26.COV2.S vaccination.
  Interventions: Biological: Ad26.COV2.S; Other: Placebo

INTERVENTIONS:
Biological: Ad26.COV2.S — Ad26.COV2.S vaccine will be administered on Day 1 and Day 57 in the double-blind phase. At unblinding visit Ad26.COV2.S vaccine will be administered to participants at Day 57 who have not yet received second vaccination and in newly enrolled participants as either single dose on Day 1 or two doses on Day 1 and Day 57. Single dose of Ad26.COV2.S vaccine will also be administered to participants initially receiving placebo. Single booster dose of Ad26.COV2.S vaccine will be given to participants in the open label phase who have received only a single vaccination with Ad26.COV2.S.
  Other Names: JNJ-78436735; Ad26COVS1; VAC31518
Other: Placebo — Placebo will be administered as IM injection on Day 1 and Day 57.
  Arms: Placebo

SUMMARY:
The study will evaluate the efficacy of Ad26.COV2.S in the prevention of molecularly confirmed moderate to severe/critical coronavirus disease-2019 (COVID-19), as compared to placebo, in SARS-CoV-2 seronegative adults in the double-blind phase and to describe COVID-19 outcomes, safety, and immunogenicity in the different study cohorts in open-label phase.

DETAILED DESCRIPTION:
The aim of the COVID-19 vaccine clinical development program is to develop a safe and effective vaccine for the prevention of COVID-19. Ad26.COV2.S, a COVID-19 vaccine based on a human replication-incompetent Ad26 vector, constructed to encode the severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) virus spike (S) protein, is being developed. The study will consist of: a screening phase (up to 28 days), study period (60-week), and a long-term follow-up period (1 additional year). The total study duration will be maximum 2 years and 3 months for the participants. Assessments for efficacy (COVID-19 signs and symptoms, etc.), immunogenicity (such as humoral immune responses), and safety (such as adverse events [AEs] monitoring) will be performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Contraceptive (birth control) use should be consistent with local regulations regarding the acceptable methods of contraception for those participating in clinical studies
* All participants of childbearing potential must: have a negative highly sensitive urine pregnancy test at screening; and have a negative highly sensitive urine pregnancy test immediately prior to each study vaccine administration
* Participant agrees to not donate bone marrow, blood, and blood products from the first study vaccine administration until 3 months after receiving the last dose of study vaccine
* Must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study
* Must be able to read, understand, and complete questionnaires in the electronic clinical outcome assessment (eCOA) (that is, the coronavirus disease-2019 [COVID 19] signs and symptoms surveillance question, the e-Diary, and the electronic patient-reported outcomes (ePROs)

Exclusion Criteria:

* Participant has a clinically significant acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature greater than or equal to (>=) 38.0 degree Celsius (100.4-degree Fahrenheit) within 24 hours prior to the planned first dose of study vaccine; randomization at a later date is permitted at the discretion of the investigator and after consultation with the sponsor
* Participant has a known or suspected allergy or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients
* Participant received or plans to receive: (a) licensed live attenuated vaccines - within 28 days before or after planned administration of study vaccine; and (b) other licensed (not live) vaccines - within 14 days before or after planned administration of study vaccine
* Participant previously received a coronavirus vaccine
* Participant received an investigational drug within 30 days (including investigational drugs for prophylaxis of COVID-19) or used an invasive investigational medical device within 30 days or received investigational immunoglobulin (Ig) or investigational monoclonal antibodies within 3 months, or received convalescent serum for COVID-19 treatment within 4 months or received an investigational vaccine (including investigational Adenoviral-vectored vaccines) within 6 months before the planned administration of the first dose of study vaccine or is currently enrolled or plans to participate in another investigational study during the course of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31835 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2023-06-18 (Actual); Study Completion 2023-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (125):
- United States (62):
  - Achieve Clinical Research, LLC, Vestavia Hills, Alabama
  - Hope Research Institute, Phoenix, Arizona
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Quality of Life Medical & Research Center, LLC, Tucson, Arizona
  - Synexus Clinical Research US Inc, Tucson, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - Synexus Clinical Research US Inc, Cerritos, California
  - eStudySite, Chula Vista, California
  - Ark Clinical Research, Long Beach, California
  - Anthony Mills Medical, Inc, Los Angeles, California
  - Benchmark Research, Sacramento, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Paradigm Clinical Research Centers, Inc., Wheat Ridge, Colorado
  - JEM Research LLC, Atlantis, Florida
  - Prestige Clinical Research Center, Inc., Coral Gables, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Health Awareness inc., Jupiter, Florida
  - Altus Research, Inc, Lake Worth, Florida
  - Compass Research, Melbourne, Melbourne, Florida
  - Suncoast Research Group, Miami, Florida
  - Behavioral Clinical Research , Inc, North Miami, Florida
  - Clinical NeuroScience Solutions Inc, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Meridien Research, St. Petersburg, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Accel Research Sites, Eatonton, Georgia
  - The University Of Chicago Medicine, Chicago, Illinois
  - Great Lakes Clinical Trials, Chicago, Illinois
  - The South Bend Clinic Center for Research, South Bend, Indiana
  - Heartland Research Associates, LLC, Newton, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Centex Studies, Inc., Lake Charles, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Centennial Medical Group, Elkridge, Maryland
  - Optimal Research, Rockville, Maryland
  - Meridian Clinical Research, LLC, Rockville, Maryland
  - Henry Ford Health Systems, Detroit, Michigan
  - Cherry Street Services, Inc., Grand Rapids, Michigan
  - Washington University School Of Medicine, St Louis, Missouri
  - Hassman Research Institute, LLC., Berlin, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Medpharmics, LLC, Albuquerque, New Mexico
  - Meridian Clinical Research, LLC, Endwell, New York
  - Regional Clinical Research, Inc., Endwell, New York
  - Allergy Asthma Immunology of Rochester, PC (AAIR) - Research Center, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - American Health Network, LLC, Charlotte, North Carolina
  - Wilmington Health Associates, Wilmington, North Carolina
  - CTI Clinical Trial and Consulting Services, Cincinnati, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Centennial Medical Center, Nashville, Tennessee
  - Centex Studies, Inc., Houston, Texas
  - Texas Center for Drug Development Inc, Houston, Texas
  - Centex Studies, Inc., McAllen, Texas
  - Endeavor Clinical Trials, LLC, San Antonio, Texas
  - Tranquility Clinical Research, Webster, Texas
  - JBR Clinical Research, Salt Lake City, Utah
  - Alliance for Multispeciality Research, Norfolk, Virginia
- Belgium (6):
  - Anima, Alken
  - Institute of Tropical Medicine Antwerp, Antwerp
  - Center for Vaccinology (CEVAC), Ghent
  - UZ Leuven, Leuven
  - Az Sint-Maarten, Mechelen
  - Private Practice RESPISOM Namur, Namur
- Brazil (5):
  - Hospital Nossa Senhora da Conceicao S A, Porto Alegre
  - Ministerio da Saude - Hospital dos Servidores do Estado - RJ, Rio de Janeiro
  - Instituto Nacional de Infectologia Evandro Chagas (INI) - FIOCRUZ, Rio de Janeiro
  - Instituto de infectologia Emilio Ribas, São Paulo
  - Centro de Referencia E Treinamento Dst/Aids, São Paulo
- Colombia (5):
  - Fundacion Cardiomet CEQUIN, Armenia
  - IPS Centro Cientifico Asisitencial Jose Luis Accini S.A.S., Barranquilla
  - Asistencia Cientifica de Alta Complejidad S.A.S, Bogotá
  - Centro Medico Imbanaco de Cali S.A., Cali
  - T Y C Inversiones S A S Grupsalud, Santa Marta
- France (8):
  - CHU de Montpellier Hopital Saint Eloi, Montpellier
  - Hopital Cochin, Paris
  - Hopital Saint-Antoine, Paris
  - Groupe Hospitalier Sud Hôpital Haut-Leveque Service d'hematologie, Pessac
  - CHU Saint Etienne Hopital Nord, Saint-Etienne
  - Hopital Rangueil, Toulouse
  - Hopital Purpan, Toulouse
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
- Klinikum rechts der Isar der TU Munchen, München, Germany
- Philippines (5):
  - Riverside Medical Center, Bacolod
  - West Visayas State University Medical Center, Iloilo City
  - Tropical Disease Foundation, Makati
  - Makati Medical Center, Manila
  - Medical Center Manila, Manila
- South Africa (8):
  - TREAD Research Tygerberg Hospital, Cape Town
  - Centre of Tuberculosis Research Innovation, Cape Town
  - Worthwhile Clinical trials, Johannesburg
  - Peermed Clinical Trial Centre, Kempton Park
  - Dr AA Mahomed Medical Centre, Moloto South
  - VX Pharma, Pretoria
  - Dr J.M. Engelbrecht Trial Site, Somerset West
  - Be Part Yoluntu Centre, Western Cape
- Spain (9):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. Quiron Barcelona, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. de La Princesa, Madrid
  - Clinica Univ. de Navarra, Madrid
  - Hosp. Univ. de La Paz, Madrid
  - Hosp. Quiron Madrid Pozuelo, Madrid
  - Clinica Univ. de Navarra, Pamplona
- United Kingdom (16):
  - Queen Elizabeth Hospital, Birmingham
  - Powys Teaching Local Health Board - Bronllys Hospital, Brecon
  - Brighton & Sussex University Hospitals NHS Trust, Brighton
  - University Hospitals Bristol NHS Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Ninewells Hospital, Dundee
  - Royal Free Hospital, Hampstead
  - Leicester Royal Infirmary, Leicester
  - Guy's and St Thomas' Hospital, London
  - Imperial College London and Imperial College Healthcare NHS Trust, London
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - University of Oxford, Oxford
  - Derriford Hospital, Plymouth
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Hardt K, Vandebosch A, Sadoff J, Le Gars M, Truyers C, Lowson D, Van Dromme I, Vingerhoets J, Kamphuis T, Scheper G, Ruiz-Guinazu J, Faust SN, Spinner CD, Schuitemaker H, Van Hoof J, Douoguih M, Struyf F; ENSEMBLE2 study group. Efficacy, safety, and immunogenicity of a booster regimen of Ad26.COV2.S vaccine against COVID-19 (ENSEMBLE2): results of a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Infect Dis. 2022 Dec;22(12):1703-1715. doi: 10.1016/S1473-3099(22)00506-0. Epub 2022 Sep 13. PMID 36113538

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 31835 participants were randomized, out of which 130 participants were randomized but not vaccinated. Hence, 31705 participants received vaccination in both double blind (DB) and open label (OL) phase. After completion of DB phases more participants were enrolled therefore, the started count of DB+OL phase is exceeding the started count for DB phase.
Pre-assignment Details: Due to change in the planned analysis, combined data of "double blind (DB)" and "open label (OL)" phase was collected and analyzed after completion of the double-blind phase. Results of safety outcome measures (OMs) were also collected and analyzed for combined DB and OL phase. Hence, safety data is reported only in adverse event section and not repeated in the OMs section.
Groups:
- Double Blind Phase: Ad26.COV2.S: Participants received a single dose of 0.5 milliliter (mL) adenovirus type 26 vector coronavirus-2 spike protein (Ad26.COV2.S) 5*10^10 viral particles (vp) vaccine intramuscularly on Day 1 and Day 57.
- Double Blind Phase: Placebo: Participants received a single dose of placebo matching to Ad26.COV2.S 5*10^10 vp vaccine intramuscularly on Day 1 and Day 57.
- Combined Double-blind and Open-label Phase: All Participants: Each participant was initially randomized to receive 1 dose of 0.5 mL Ad26.COV2.S 5*10^10 vp vaccine intramuscularly on Day 1 and on Day 57 or 1 dose of placebo vaccine intramuscularly on Day 1 and on Day 57 during the DB phase (up to 7.2 months). Following authorization of COVID-19 vaccine(s) in their country, participants could request to be unblinded to receive a different authorized/licensed COVID-19 vaccine outside of the study at any time during the study. Following Emergency Use Authorization of Ad26.COV2.S in the United States, all participants were unblinded and entered OL phase, and those participants that received placebo could receive a single dose of Ad26.COV2.S 5*10^10 vp vaccine. Later it was allowed to have a booster vaccination with a single dose of Ad26.COV2.S 5*10^10 vp vaccine for those participants that received a single dose of Ad26.COV2.S vaccine in the study.
Period: DB Phase (Day 1 up to 7.2 Months)
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo | Combined Double-blind and Open-label Phase: All Participants
Started | 15708 | 15592 | 0
FAS Post-Dose 1 Population (7 participants (3 in the Ad26 group, 4 in the placebo group) received a COVID-19 vaccination outside of the study prior to first study vaccination. These participants were excluded from post-dose 1 FAS.) | 15705 | 15588 | 0
Non-FAS Post-Dose 1 Population (Participants who received a COVID-19 vaccination outside of the study prior to first study vaccination.) | 3 | 4 | 0
FAS Post-Dose 1 Safety Subset (Subset of FAS) | 3015 | 3052 | 0
Non-FAS Post-Dose 1 Safety Subset (Subset of FAS) | 1 | 0 | 0
Completed | 15007 | 13834 | 0
Not Completed | 701 | 1758 | 0
Not completed — Adverse Event | 5 | 10 | 0
Not completed — Death | 6 | 13 | 0
Not completed — Lost to Follow-up | 170 | 219 | 0
Not completed — Physician Decision | 15 | 6 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 7 | 0
Not completed — Withdrawal by Subject | 468 | 1273 | 0
Not completed — Initiated Prohibited Medication | 10 | 75 | 0
Not completed — Rolled Over into Different Clinical Trial | 0 | 3 | 0
Not completed — Technical Problems | 0 | 2 | 0
Not completed — Other | 26 | 149 | 0
Period: DB + Open-label Phase (2 Years 6 Months)
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo | Combined Double-blind and Open-label Phase: All Participants
Started | 0 | 0 | 31705 (Participants of DB phase that entered into the OL phase. After completion of DB phases more participants were enrolled therefore, the started count of DB+OL phase is exceeding the started count for DB phase.)
Completed | 0 | 0 | 21018
Not Completed | 0 | 0 | 10687
Not completed — Adverse Event | 0 | 0 | 14
Not completed — Death | 0 | 0 | 131
Not completed — Lost to Follow-up | 0 | 0 | 3796
Not completed — Physician Decision | 0 | 0 | 178
Not completed — Pregnancy | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 5922
Not completed — Initiated Prohibited Medication | 0 | 0 | 92
Not completed — Rolled Over into Different Clinical Trial | 0 | 0 | 48
Not completed — Technical Problems | 0 | 0 | 17
Not completed — Sponsor Decision | 0 | 0 | 1
Not completed — Other | 0 | 0 | 477

BASELINE CHARACTERISTICS:
Population: All Participants arm included combined baseline data for DB and OL phase as per change in the planned analysis.
Arm/Group | Combined Double-blind and Open-label Phase: All Participants
Number analyzed (Participants) | 31705
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (14.46)
Age, Customized [Count of Participants; unit: Participants]
  From 18 to 64 years | 25993
  From 65 to 84 years | 5640
  85 years and over | 72
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 15032
  Male | 16669
  Undifferentiated | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    American Indian or Alaska Native | 798
    Asian | 2806
    Black or African American | 2677
    Native Hawaiian or Other Pacific Islander | 78
    White | 24074
    More Than One Race | 460
    Unknown or Not Reported | 812
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 5799
    Not Hispanic or Latino | 25011
    Unknown or Not Reported | 895
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 2981
  BRAZIL | 500
  COLOMBIA | 2149
  FRANCE | 714
  GERMANY | 100
  PHILIPPINES | 1572
  SOUTH AFRICA | 2073
  SPAIN | 3132
  UNITED KINGDOM | 5905
  UNITED STATES | 12579

OUTCOME MEASURES:

1. Primary Outcome: Double Blind Phase: Number of Participants With First Occurrence of Molecularly Confirmed Moderate to Severe/Critical COVID-19 in Seronegative Participants With Onset at Least 14 Days After the Second Vaccination
Description: Molecularly confirmed moderate to severe/critical COVID-19 was defined as a severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) positive reverse transcription/polymerase chain reaction (RT-PCR) or molecular test result from any available respiratory tract sample (example, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample. Moderate included one sign or symptom such as respiratory rate >=20 breaths per minute (min) and symptoms such as shortness of breath or two signs or symptoms such as heart rate >=90 beats/min and symptoms such as cough from a list of signs and symptoms and severe/critical included one of the following signs and symptoms: respiratory rate >=30 breaths/min, heart rate >=125 beats/min, oxygen saturation (SpO2) <=93 percent (%) on room air at sea level respiratory failure, evidence of shock, significant acute renal, hepatic, or neurologic dysfunction, admission to Intensive Care Unit (ICU), death defined as per FDA guidance.
Time Frame: From at least 14 days after second vaccination on Day 57 (Day 71) up to end of double blind phase (7.2 months)
Population: Per-protocol efficacy (PP) set: participants in FAS who received 2 doses of DB study vaccine, were PCR negative at time of first vaccination, were seronegative at time of first vaccination and at 14 days after second vaccination and had no other major protocol deviations to possibly impact efficacy of vaccine before unblinding. Participants who had a positive PCR test between Day 1 and Day 70 and participants who discontinued prior to 14 days post-dose 2 were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 6024 | 5615
Participants | 14 | 52

2. Secondary Outcome: Double Blind Phase: Number of Participants With First Occurrence of Molecularly Confirmed Moderate to Severe/Critical COVID-19 Regardless of Serostatus With Onset At Least 1 Day After the First Day 1 Vaccination
Description: Molecularly confirmed moderate to severe/critical COVID-19 was defined as a SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (example, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample. Moderate included one sign or symptom such as respiratory rate greater than or equal to (>=) 20 breaths per minute and symptoms such as shortness of breath or two signs or symptoms such as heart rate >= 90 beats per min and symptoms such as cough from a list of signs and symptoms and severe/critical included one of the following signs and symptoms: respiratory rate >=30 breaths/minute, heart rate >=125 beats/minute, SpO2 less than or equal to (<=) 93% on room air at sea level respiratory failure, evidence of shock, significant acute renal, hepatic, or neurologic dysfunction, admission to the ICU, death defined as per US Food and Drug Administration (FDA) guidance.
Time Frame: From at least 1 day after first vaccination on Day 1 (Day 2) up to end of double blind phase (7.2 months)
Population: Full analysis set (FAS) included all randomized participants with at least 1 documented study vaccine administration, regardless of protocol deviations and serostatus at enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 15708 | 15592
Participants | 115 | 259

3. Secondary Outcome: Double Blind Phase: Number of Participants With First Occurrence of Molecularly Confirmed Moderate to Severe/Critical COVID-19 Regardless of Serostatus With Onset at Least 14 Days After the Second Vaccination
Description: Molecularly confirmed moderate to severe/critical COVID-19 was defined as a SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (example, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample. Moderate included one sign or symptom such as respiratory rate >= 20 breaths per minute and symptoms such as shortness of breath or two signs or symptoms such as heart rate >= 90 beats per min and symptoms such as cough from a list of signs and symptoms and severe/critical included one of the following signs and symptoms: respiratory rate >=30 breaths/minute, heart rate >=125 beats/minute, SpO2 <= 93% on room air at sea level respiratory failure, evidence of shock, significant acute renal, hepatic, or neurologic dysfunction, admission to the ICU, death defined as per FDA guidance.
Time Frame: From at least 14 days after second vaccination on Day 57 (Day 71) up to end of double blind phase (7.2 months)
Population: PP set: included participants of the FAS who received 2 doses of DB study vaccine, regardless of their serostatus at time of first vaccination and at 14 days after second vaccination, were PCR negative at time of first vaccination and had no other major protocol deviations to possibly impact efficacy of vaccine before unblinding. Participants who had a positive PCR test between Day 1 and Day 70 and participants who discontinued prior to 14 days post-dose 2 were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 6813 | 6370
Participants | 14 | 53

4. Secondary Outcome: Double Blind Phase: Number of Participants With First Occurrence of Molecularly Confirmed Moderate to Severe/Critical COVID-19 in Seronegative Participants With Onset at Least 1 Day After the First Day 1 Vaccination
Description: as for outcome 3
Time Frame: From at least 1 day after first vaccination on Day 1 (Day 2) up to end of double blind phase (7.2 months)
Population: Full analysis seronegative set included all randomized participants with at least 1 documented study vaccine administration, regardless of protocol deviations and who were seronegative at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 13951 | 13871
Participants | 112 | 256

5. Secondary Outcome: Double Blind Phase: Number of Participants With First Occurrence of Molecularly Confirmed Moderate to Severe/Critical COVID-19 With Onset at Least 14 Days After the First Day 1 Vaccination
Description: as for outcome 3
Time Frame: From at least 14 days after first vaccination on Day 1 (Day 15) up to end of double blind phase (7.2 months)
Population: Per-protocol first dose efficacy (PPFD) population: Participants in FAS who received at least first dose of study vaccine in the double-blind phase and who were PCR negative at the time of first vaccination, who were not seropositive at baseline and who had no major protocol deviations before unblinding that were judged to possibly impact the efficacy of the vaccine. Participants who had a positive PCR test between Days 1 and 14 and participants who discontinued prior to Day 15 were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 13316 | 13286
Participants | 72 | 216

6. Secondary Outcome: Double Blind Phase: Number of Participants With First Occurrence of Molecularly Confirmed Moderate to Severe/Critical COVID-19 With Onset at Least 28 Days After the First Day 1 Vaccination
Description: as for outcome 3
Time Frame: From at least 28 days after the first vaccination on Day 1 (Day 29) up to end of double blind phase (7.2 months)
Population: PPFD population: Participants in FAS who received at least first dose of study vaccine in the double-blind phase and who were PCR negative at the time of first vaccination, who were not seropositive at baseline and who had no major protocol deviations before unblinding that were judged to possibly impact the efficacy of the vaccine. Participants who had a positive PCR test between Day 1 and Day 28 and participants who discontinued prior to Day 29 were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 12632 | 12402
Participants | 52 | 161

7. Secondary Outcome: Double Blind Phase: Number of Participants With First Occurrence of COVID-19 Requiring Medical Intervention With Onset at Least 14 Days After the Second Vaccination
Description: Number of participants with first occurrence of COVID-19 requiring medical intervention (such as a composite endpoint of hospitalization, ICU admission, mechanical ventilation, and extracorporeal membrane oxygenation [ECMO]), linked to objective measures such as decreased oxygenation, X-ray or computed tomography [CT] findings and linked to any molecularly confirmed, COVID-19 with onset at least 14 days post second vaccination were reported.
Time Frame: From at least 14 days after second vaccination on Day 57 (Day 71) up to end of double blind phase (7.2 months)
Population: PP set: participants in FAS who received 2 doses of DB study vaccine, were PCR negative at time of first vaccination, were seronegative at time of first vaccination and at 14 days after second vaccination and had no other major protocol deviations to possibly impact efficacy of vaccine before unblinding. Participants who had a positive PCR test between Day 1 and Day 70 and participants who discontinued prior to 14 days post-dose 2 were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 6024 | 5615
Participants | 0 | 5

8. Secondary Outcome: Double Blind Phase: Area Under the Curve (AUC) of SARS-CoV-2 Viral Load as Assessed by Quantitative RT-PCR in Participants With Molecularly Confirmed Symptomatic COVID-19 With Onset at Least 14 Days After Second Vaccination
Description: AUC of SARS-CoV-2 viral load was assessed in confirmed COVID-19 cases using RT-PCR. Nasal swabs were used to detect and/or quantify SARS-CoV-2. Due to change in the planned analysis, data was collected and analyzed for participants with molecularly confirmed symptomatic COVID-19 regardless of severity that is mild, moderate or severe and was not collected and analyzed separately for moderate to severe cases.
Time Frame: From Day 71 up to end of the COVID-19 episode (up to 90 days)
Population: PP set: participants in FAS who received 2 doses of double-blind study vaccine, were PCR negative at the time of first vaccination, were seronegative at the time of first vaccination and at 14 days after second vaccination and had no other major protocol deviations to possibly impact efficacy of vaccine before unblinding. 'N' (overall number of participants analyzed) = participants evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: Log10 copies*day per milliliter
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 11 | 47
Log10 copies*day per milliliter | 847.68 (242.375) | 1023.59 (156.298)

9. Secondary Outcome: Double Blind Phase: Number of Participants With First Occurrence of Molecularly Confirmed Mild COVID-19 With Onset at Least 14 Days After the Second Vaccination
Description: Molecularly confirmed mild Covid-19 was defined as a SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (example, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample and one of the following signs and symptoms: fever (>=38 degree Celsius or >=100.4 degree Fahrenheit), sore throat, malaise (loss of appetite, generally unwell, fatigue, physical weakness), headache, muscle pain (myalgia), gastrointestinal symptoms, cough, chest congestion, runny nose, wheezing, skin rash, eye irritation or discharge, chills, new or changing olfactory or taste disorders, red or bruised looking feet or toes, or shaking chills or rigors.
Time Frame: From at least 14 days after second vaccination on Day 57 (Day 71) up to end of double blind phase (7.2 months)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 6024 | 5615
Participants | 0 | 1

10. Secondary Outcome: Double Blind Phase: Number of Participants With First Occurrence of Molecularly Confirmed COVID-19 Defined by the US FDA Harmonized Case Definition With Onset at Least 14 Days After the Second Vaccination
Description: Molecularly confirmed COVID-19 was defined as SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (example, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample; and COVID-19 symptoms consistent with those defined by the US FDA harmonized case definition at the time of finalization of the study protocol: fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, and diarrhea.
Time Frame: From at least 14 days after second vaccination on Day 57 (Day 71) up to end of double blind phase (7.2 months)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 6024 | 5615
Participants | 12 | 52

11. Secondary Outcome: Double Blind Phase: Number of Participants With Burden of Disease (BOD) Based on First Occurrence of Molecularly Confirmed Symptomatic COVID-19 With Onset at Least 14 Days After the Second Vaccination
Description: BOD is a weighted version of the mild, moderate, and severe/critical vaccine efficacies and was evaluated based on the first occurrence of molecularly confirmed COVID-19, including mild, moderate or severe/critical COVID-19 case.
Time Frame: From at least 14 days after second vaccination on Day 57 (Day 71) up to end of double blind phase (7.2 months)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 6024 | 5615
Participants | 14 | 53

12. Secondary Outcome: Double Blind Phase: Number of Participants With Serologic Conversion Between Day 71 up to Unblinding Visit Using an Enzyme-linked Immunosorbent Assay (ELISA)
Description: Number of participants with serologic conversion between Day 71 up to unblinding visit using an ELISA were reported. Due to change in planned analysis, data was collected and analyzed between Day 71 up to unblinding visit instead of from baseline to unblinding visit.
Time Frame: From Day 71 up to unblinding visit (7.2 months)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 6024 | 5615
Participants | 32 | 45

13. Secondary Outcome: Double Blind Phase: Number of Participants With Asymptomatic Infection Detected By Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) With Onset at Least 14 Days After the Second Vaccination
Description: Number of participants with asymptomatic infection detected by RT-PCR with onset at least 14 days after the second vaccination (Day 71) were reported.
Time Frame: From at least 14 days after second vaccination on Day 57 (Day 71) up to end of double blind phase (7.2 months)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 6024 | 5615
Participants | 40 | 56

14. Secondary Outcome: Double Blind Phase: Number of Participants With First Occurrence of SARS-CoV-2 Infection (Serologically and/or Molecularly Confirmed) With Onset at Least 14 Days After the Second Vaccination
Description: Number of participants with first occurrence of SARS-CoV-2 infection (serologically and/or molecularly confirmed) with onset at least 14 days after the second vaccination (Day 71) were reported.
Time Frame: From at least 14 days after second vaccination on Day 57 (Day 71) up to end of double blind phase (7.2 months)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 6024 | 5615
Participants | 60 | 113

15. Secondary Outcome: Double Blind Phase: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product that does not necessarily have a causal relationship with the vaccine. SAE was any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: From Day 1 up to end of double blind phase (7.2 months)
Population: FAS post dose 1 population included FAS participants excluding the participants who received a COVID-19 vaccination outside of the study prior to first study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 15705 | 15588
Participants | 104 | 136

16. Secondary Outcome: Double Blind Phase: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: Number of participants with AESIs were reported. AESIs were significant AEs that were judged to be of special interest because of clinical importance, known or suspected class effects, or based on nonclinical signals. Thrombosis with Thrombocytopenia Syndrome (TTS), a syndrome characterized by a combination of both a thrombotic event and thrombocytopenia, was considered to be an AESI in this study. A suspected TTS case was defined as: Thrombotic events: suspected deep vessel venous or arterial thrombotic events; Thrombocytopenia, defined as platelet count below 150,000/micro liter.
Time Frame: From Day 1 up to end of double blind phase (7.2 months)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 15705 | 15588
Participants | 2 | 1

17. Secondary Outcome: Double Blind Phase: Number of Participants With Medically-Attended Adverse Events (MAAEs)
Description: An AE was any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product that does not necessarily have a causal relationship with the vaccine. MAAEs were defined as AEs with medically-attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason.
Time Frame: From Day 1 up to 7.2 months
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 15705 | 15588
Participants | 1033 | 1003

18. Secondary Outcome: Double-Blind: Number of Participants With MAAEs Leading to Study Discontinuation
Description: as for outcome 17
Time Frame: From Day 1 up to end of double blind phase (7.2 months)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 15705 | 15588
Participants | 4 | 8

19. Secondary Outcome: Double Blind Phase: Number of Participants With Solicited Local Adverse Events (AEs) During 7 Days Following Each Vaccination
Description: An AE was any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product that does not necessarily have a causal relationship with the vaccine. Participants who were enrolled in safety subset (SS) were asked to note in the e-Diary occurrences of injection site pain/tenderness, erythema, and swelling at the study vaccine injection site daily for 7 days post each vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days after first vaccination on Day 1 (up to Day 8), 7 days after second vaccination on Day 57 (up to Day 64)
Population: Safety population was a subset of FAS for analyzing solicited local AEs. 'N' (overall number of participants analyzed) = participants evaluable for this outcome; 'n' (number analyzed) = participants evaluable at specific time points. N=0 in 'DB: Non-FAS Post-Dose 1: Placebo' arm, as no participant was evaluable in the FAS subset of this arm. n=0 in 'DB: Non-FAS Post-Dose 1' arm signifies the time point was not applicable since the participant did not receive a second vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Double Blind Phase: Non-FAS Post-Dose 1: Ad26.COV2.S: Participants who received a COVID-19 vaccination outside of the study prior to first study vaccination were randomized to receive a single dose of 0.5 mL Ad26.COV2.S 5*10^10 vp vaccine intramuscularly on Day 1.
- Double Blind Phase: Non-FAS Post-Dose 1: Placebo: Participants who received a COVID-19 vaccination outside of the study prior to first study vaccination were randomized to receive a single dose of placebo matching to Ad26.COV2.S 5*10^10 vp vaccine intramuscularly on Day 1.
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo | Double Blind Phase: Non-FAS Post-Dose 1: Ad26.COV2.S | Double Blind Phase: Non-FAS Post-Dose 1: Placebo
Number analyzed (Participants) | 3015 | 3052 | 1 | 0
Participants
  Day 8 | 1676 | 653 | 1 |
  Day 64: number analyzed (Participants) | 1559 | 1425 | 0 | 0
  Day 64 | 896 | 252 |  |

20. Secondary Outcome: Double Blind Phase: Number of Participants With Solicited Systemic AEs During 7 Days Following Each Vaccination
Description: An AE was any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product that does not necessarily have a causal relationship with the vaccine. Participants who were enrolled in safety subset were instructed on how to record daily temperature using a thermometer provided for home use. Participants recorded temperature in e-Diary in evening of the day of vaccination, and then daily for next 7 days approximately at same time each day. If more than 1 measurement was made on any given day, the highest temperature of that day was recorded in e-Diary. Fever was defined as endogenous elevation of body temperature >= 38.0 degree Celsius or >=100.4-degree Fahrenheit, as recorded in at least 1 measurement. Participants also noted the signs and symptoms in e-Diary on a daily basis for 7 days post each vaccination (day of vaccination and subsequent 7 days), for the following events: fatigue, headache, nausea, myalgia.
Time Frame: 7 days after first vaccination on Day 1 (up to Day 8), 7 days after second vaccination on Day 57 (up to Day 64)
Population: Safety population was subset of FAS for analysis of solicited systemic AEs. 'N' (overall number of participants analyzed)=participants evaluable for this outcome measure; 'n' (number analyzed)= participants evaluable at specified time points. N=0 in 'DB: Non-FAS Post-Dose 1: Placebo' arm, as no participant was evaluable in the FAS subset of this arm. n=0 in 'DB: Non-FAS Post-Dose 1' arm signifies the time point was not applicable since the participant did not receive a second vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo | Double Blind Phase: Non-FAS Post-Dose 1: Ad26.COV2.S | Double Blind Phase: Non-FAS Post-Dose 1: Placebo
Number analyzed (Participants) | 3015 | 3052 | 1 | 0
Participants
  Day 8 | 1764 | 1138 | 1 |
  Day 64: number analyzed (Participants) | 1559 | 1425 | 0 | 0
  Day 64 | 821 | 442 |  |

21. Secondary Outcome: Double Blind Phase: Number of Participants With Unsolicited Adverse Events (AEs) During 28 Days Post Each Vaccination
Description: An AE was any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product that does not necessarily have a causal relationship with the vaccine. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days after first vaccination on Day 1 (up to Day 29), 28 days after second vaccination on Day 57 (up to Day 85)
Population: Safety population was subset of FAS for analysis of unsolicited AEs. 'N' (overall number of participants analyzed) = participants evaluable for this outcome measure; 'n' (number analyzed) = participants evaluable at specified time points. N=0 in 'DB: Non-FAS Post-Dose 1: Placebo' arm, as no participant was evaluable in the FAS subset of this arm. n=0 in 'DB: Non-FAS Post-Dose 1' arm signifies the time point was not applicable since the participant did not receive a second vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo | Double Blind Phase: Non-FAS Post-Dose 1: Ad26.COV2.S | Double Blind Phase: Non-FAS Post-Dose 1: Placebo
Number analyzed (Participants) | 3015 | 3052 | 1 | 0
Participants
  Day 29 | 454 | 332 | 0 |
  Day 85: number analyzed (Participants) | 1559 | 1425 | 0 | 0
  Day 85 | 159 | 120 |  |

22. Secondary Outcome: Double Blind Phase: SARS-CoV-2 Binding Antibodies Assessed by ELISA
Description: Binding antibodies to SARS-CoV-2 S protein as assessed by ELISA to measure humoral immune response was reported. The lower limit of quantification (LLOQ) was 50.3 ELISA units per milliliter (EU/mL). A sample was considered positive if the value was strictly greater than the LLOQ (>LLOQ).
Time Frame: At Baseline (Day 1), Days 29, 57 and 71
Population: Per protocol immunogenicity (PPI) set: all randomized and vaccinated participants (received both vaccines in DB phase, including those who were part of immunogenicity subset and for whom immunogenicity data were available, excluding participants with major protocol deviations expected to impact immunogenicity outcomes. N (overall number of participants analyzed) = participants evaluated for this outcome measure, n (number analyzed) = number of participants evaluable at specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Unit/milliliter (EU/mL)
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo
Number analyzed (Participants) | 157 | 149
ELISA Unit/milliliter (EU/mL)
  Day 1 | NA [NA to NA] — Geometric mean and 95% confidence interval could not be estimated as the analyzed values were below the LLOQ (50.3 EU/mL). | NA [NA to NA] — Geometric mean and 95% confidence interval could not be estimated as the analyzed values were below the LLOQ (50.3 EU/mL).
  Day 29: number analyzed (Participants) | 140 | 124
  Day 29 | 367 [295 to 456] | NA [NA to NA] — Geometric mean and 95% confidence interval could not be estimated as the analyzed values were below the LLOQ (50.3 EU/mL).
  Day 57: number analyzed (Participants) | 150 | 111
  Day 57 | 518 [422 to 635] | NA [NA to NA] — Geometric mean and 95% confidence interval could not be estimated as the analyzed values were below the LLOQ (50.3 EU/mL).
  Day 71: number analyzed (Participants) | 78 | 62
  Day 71 | 2220 [1794 to 2748] | NA [NA to NA] — Geometric mean and 95% confidence interval could not be estimated as the analyzed values were below the LLOQ (50.3 EU/mL).

ADVERSE EVENTS:
Time Frame: DB phase: All-cause mortality and SAEs: From Day 1 till end of DB phase (up to 7.2 months), Solicited AEs: 7 days after first vaccination on Day 1 (up to Day 8), 7 days after second vaccination on Day 57 (up to Day 64) ; All participants arm: All-cause mortality and SAEs: Day 1 up to end of study (up to 2 years 6 months); DB Phase: Other AEs: 28 days after first vaccination on Day 1 (up to Day 29 ), 28 days after vaccination 2 on Day 57 (up to Day 85)
Description: All-cause mortality/SAE: Per change in planned analysis, due to complex vaccination schedules, combined data for DB and OL was analyzed in the 'All Participant' arm after unblinding. As pre-specified: (a) only deaths/SAEs were planned to be collected in OL phase, (b) safety subset of FAS was used to analyze other AEs in DB phase. At risk=0 for 'All Participant' arm for other AEs as data for other AEs was not collected after unblinding (end of DB phase) per planned analysis. DB: MedDRA v24.0.
Arm/Group | Double Blind Phase: Ad26.COV2.S | Double Blind Phase: Placebo | Combined Double-blind and Open-label Phase: All Participants | Double Blind Phase: Non-FAS Post-Dose 1: Ad26.COV2.S | Double Blind Phase: Non-FAS Post-Dose 1: Placebo
All-Cause Mortality (participants affected / at risk) | 6/15705 | 13/15588 | 131/31705 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 104/15705 | 136/15588 | 1583/31705 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 2234/3015 | 1531/3052 | 0/0 | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind Phase: Ad26.COV2.S (N=15705) | Double Blind Phase: Placebo (N=15588) | Combined Double-blind and Open-label Phase: All Participants (N=31705) | Double Blind Phase: Non-FAS Post-Dose 1: Ad26.COV2.S (N=3) | Double Blind Phase: Non-FAS Post-Dose 1: Placebo (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 10 | 0 | 0
Anaemia megaloblastic (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0
Myelosuppression (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 18 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1 | 36 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 0 | 14 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 1 | 7 | 0 | 0
Aortic valve disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 3 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 3 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 5 | 0 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 27 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 5 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 3 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 5 | 0 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 2 | 8 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 12 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cor pulmonale (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 18 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 11 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Heart valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Microvascular coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Mitral valve disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 2 | 0 | 0
Myocardial fibrosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 4 | 24 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 3 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 1 | 4 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 4 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 2 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 3 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 4 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Brugada syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Congenital tracheomalacia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Laryngocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 5 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Basedow's disease (Endocrine disorders) | 0 | 0 | 2 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Parathyroid disorder (Endocrine disorders) | 0 | 0 | 2 | 0 | 0
Thyroid cyst (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Thyroiditis acute (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Blindness transient (Eye disorders) | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 5 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 2 | 0 | 0
Epiretinal membrane (Eye disorders) | 0 | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 2 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 3 | 0 | 0
Retinal ischaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Scleritis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 6 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Appendicitis noninfective (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Enterocele (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Epiploic appendagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Femoral hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 8 | 0 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 6 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 2 | 16 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 5 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal prolapse (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Intestinal strangulation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Lumbar hernia (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0
Mesenteric panniculitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Obstructive defaecation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 7 | 0 | 0
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Peritoneal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Retroperitoneal mass (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Salivary gland mass (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Tongue haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 7 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Volvulus of small bowel (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0
Accidental death (General disorders) | 0 | 0 | 1 | 0 | 0
Capsular contracture associated with implant (General disorders) | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 2 | 8 | 0 | 0
Death (General disorders) | 1 | 0 | 19 | 0 | 0
Death neonatal (General disorders) | 0 | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0
Hernia pain (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 6 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 4 | 0 | 0
Sudden death (General disorders) | 0 | 1 | 2 | 0 | 0
Vaccination site pain (General disorders) | 1 | 0 | 1 | 0 | 0
Vascular stent stenosis (General disorders) | 0 | 1 | 2 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 3 | 0 | 0
Biliary cyst (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 1 | 10 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 8 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 3 | 19 | 0 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Gallbladder polyp (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Gallbladder rupture (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 4 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hydrocholecystis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 2 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 2 | 0 | 0
Allergy to vaccine (Immune system disorders) | 1 | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 2 | 0 | 0
Food allergy (Immune system disorders) | 1 | 0 | 1 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Abscess jaw (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Appendiceal abscess (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 3 | 4 | 34 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Arboviral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Aspergilloma (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bartholinitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Burn infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 5 | 24 | 78 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 3 | 13 | 45 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 1 | 15 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Chronic hepatitis B (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Colonic abscess (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Complicated appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 3 | 0 | 0
Diabetic foot infection (Infections and infestations) | 0 | 1 | 2 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 7 | 0 | 0
Diverticulitis intestinal perforated (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Escherichia pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Eye infection intraocular (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 1 | 2 | 0 | 0
Gastric ulcer helicobacter (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastritis helminthic (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 5 | 0 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1 | 0 | 0
HIV infection (Infections and infestations) | 0 | 0 | 3 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Infected bite (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Lung abscess (Infections and infestations) | 1 | 1 | 2 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Meningoencephalitis herpetic (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Murine typhus (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Neurosyphilis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Plasmodium falciparum infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 45 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 5 | 0 | 0
Post-acute COVID-19 syndrome (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 6 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 4 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 22 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Shunt infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Spontaneous bacterial peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Submandibular abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Systemic candida (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Tubo-ovarian abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 14 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 10 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Wound sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 8 | 0 | 0
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Bone graft lysis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Burns third degree (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 6 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 5 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 7 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Frostbite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 6 | 0 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 5 | 0 | 0
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 5 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 3 | 0 | 0
Lisfranc fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 2 | 4 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 2 | 0 | 4 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Osteoradionecrosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 4 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 7 | 0 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 7 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1 | 12 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Snake bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 9 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0
Traumatic arthrosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 4 | 0 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 4 | 0 | 0
Biopsy liver (Investigations) | 0 | 0 | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1 | 0 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 0 | 1 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 1 | 0 | 0
Myocardial necrosis marker increased (Investigations) | 1 | 0 | 1 | 0 | 0
Sleep study (Investigations) | 0 | 0 | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 1 | 0 | 0
Adult failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 8 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 4 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 6 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 5 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 0 | 0
Chondrolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 9 | 0 | 0
Infrapatellar fat pad inflammation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 1 | 16 | 0 | 0
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Meniscopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 70 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 8 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Vertebral lateral recess stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 8 | 0 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Anal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4 | 0 | 0
Benign neoplasm of testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Borderline serous tumour of ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 22 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 8 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Endometrial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Follicular lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 7 | 0 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3 | 0 | 0
Lung adenocarcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 6 | 0 | 0
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 0 | 0
Malignant melanoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Oesophageal adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 0 | 0
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Osteosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Paget's disease of nipple (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Phyllodes tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 29 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 0 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Tumour of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 8 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Bell's palsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 1 | 3 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebellar stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebral amyloid angiopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 3 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 8 | 0 | 0
Cerebral thrombosis (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 1 | 12 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Diabetic ketoacidotic hyperglycaemic coma (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Facial paresis (Nervous system disorders) | 1 | 0 | 2 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 3 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 3 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 4 | 0 | 0
Hashimoto's encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 4 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hypoglossal nerve paresis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Intracranial mass (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 1 | 12 | 0 | 0
Lacunar stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 3 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 3 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 3 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Myelitis transverse (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 2 | 0 | 0
Neuromyopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Paresis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Post-traumatic epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 3 | 0 | 0
Primary headache associated with sexual activity (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Pseudostroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
SUNCT syndrome (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 8 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 4 | 0 | 0
Spinal claudication (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 11 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Thalamic infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Transient global amnesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 14 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 9 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 1 | 0 | 0
Device failure (Product Issues) | 0 | 0 | 2 | 0 | 0
Prosthetic cardiac valve malfunction (Product Issues) | 0 | 0 | 1 | 0 | 0
Acute psychosis (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 4 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 2 | 0 | 3 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 3 | 0 | 0
Conversion disorder (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 10 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Drug abuse (Psychiatric disorders) | 1 | 0 | 2 | 0 | 0
Gender dysphoria (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Nicotine dependence (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0 | 3 | 0 | 0
Psychiatric decompensation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Schizoaffective disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Schizoaffective disorder bipolar type (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 7 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 10 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 2 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 0
End stage renal disease (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 2 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 3 | 15 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 3 | 0 | 0
Renal mass (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urate nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 5 | 0 | 0
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 2 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0
Adnexal torsion (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 5 | 0 | 0
Breast discomfort (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0
Breast enlargement (Reproductive system and breast disorders) | 0 | 0 | 3 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Colpocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 5 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 3 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 7 | 0 | 0
Ovarian disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Pelvic fluid collection (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0
Vulvar dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 12 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 10 | 0 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Neonatal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pharyngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 35 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Bereavement (Social circumstances) | 0 | 1 | 1 | 0 | 0
Homicide (Social circumstances) | 0 | 1 | 1 | 0 | 0
Miscarriage of partner (Social circumstances) | 0 | 0 | 1 | 0 | 0
Aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Aneurysm thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 2 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Aortic dilatation (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 5 | 0 | 0
Aortic thrombosis (Vascular disorders) | 0 | 0 | 2 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 4 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 9 | 0 | 0
Essential hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 5 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Hypertensive urgency (Vascular disorders) | 0 | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 3 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 2 | 0 | 0
Iliac artery stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Intermittent claudication (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Malignant hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Microscopic polyangiitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Penetrating aortic ulcer (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 2 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 2 | 0 | 0
Peripheral embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Systolic hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 2 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 2 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 2 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0
Unevaluable event (General disorders) | 0 | 1 | 0 | 0 | 0
Postoperative abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind Phase: Ad26.COV2.S (N=3015) | Double Blind Phase: Placebo (N=3052) | Combined Double-blind and Open-label Phase: All Participants (N=0) | Double Blind Phase: Non-FAS Post-Dose 1: Ad26.COV2.S (N=1) | Double Blind Phase: Non-FAS Post-Dose 1: Placebo (N=0)
Nausea(Solicited) (Gastrointestinal disorders) | 666 | 387 | 0 | 0 | 0 — MedDRA version 24.0 was used for solicited non-SAEs.
Fatigue(Solicited) (General disorders) | 1531 | 897 | 0 | 0 | 0 — MedDRA version 24.0 was used for solicited non-SAEs.
Pyrexia(Solicited) (General disorders) | 177 | 18 | 0 | 0 | 0 — MedDRA version 24.0 was used for solicited non-SAEs.
Vaccination site erythema(Solicited) (General disorders) | 311 | 170 | 0 | 1 | 0 — MedDRA version 24.0 was used for solicited non-SAEs.
Vaccination site pain (General disorders) | 72 | 23 | 0 | 0 | 0
Vaccination site pain(Solicited) (General disorders) | 1818 | 664 | 0 | 1 | 0 — MedDRA version 24.0 was used for solicited non-SAEs.
Vaccination site swelling(Solicited) (General disorders) | 215 | 65 | 0 | 0 | 0 — MedDRA version 24.0 was used for solicited non-SAEs.
Myalgia(Solicited) (Musculoskeletal and connective tissue disorders) | 1346 | 572 | 0 | 1 | 0 — MedDRA version 24.0 was used for solicited non-SAEs.
Headache(Solicited) (Nervous system disorders) | 1432 | 873 | 0 | 0 | 0 — MedDRA version 24.0 was used for solicited non-SAEs.
Fatigue (General disorders) | 128 | 119 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 99 | 86 | 0 | 0 | 0
Headache (Nervous system disorders) | 138 | 120 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Per change in planned analysis, safety results for Open-label (OL) phase were included in the All Participants arm in AE section, hence are not repeated in OM section. There was no planned cross-over, the various complex vaccination sequences were a result of ethically allowing placebo participants to unblind themselves and receive active vaccination in OL phase. Hence data could not be analyzed separately for OL phase and was combined with DB phase after unblinding in 'All Participants' arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/48/NCT04614948/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT04614948/SAP_001.pdf